CLINICAL TRIAL: NCT06246916
Title: A Phase 3 Study of Fixed Dose Combinations of Fianlimab and Cemiplimab Versus Relatlimab and Nivolumab in Participants With Unresectable or Metastatic Melanoma
Brief Title: A Study With Combinations of Anti-LAG-3 and Anti-PD-1 Antibodies in Adult Participants With Advanced or Metastatic Melanoma (Harmony Head-to-Head)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3767-ONC-22122
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: Unresectable Melanoma; Metastatic Melanoma; Advanced Melanoma; Stage III; Stage IV
MeSH Terms: conditions — Melanoma | interventions — cemiplimab; Opdualag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- fianlimab+cemiplimab (Experimental): Randomized 1:1
  Interventions: Drug: fianlimab; Drug: cemiplimab
- relatlimab+nivolumab (Active Comparator): Randomized 1:1
  Interventions: Drug: relatlimab+nivolumab

INTERVENTIONS:
Drug: fianlimab — Intravenous (IV) administration every 3 weeks (Q3W) in combination with cemiplimab
  Other Names: REGN3767
  Arms: fianlimab+cemiplimab
Drug: cemiplimab — IV administration Q3W in combination with fianlimab
  Other Names: REGN2810; LIBTAYO®
  Arms: fianlimab+cemiplimab
Drug: relatlimab+nivolumab — IV administration every 4 weeks (Q4W)
  Other Names: Opdualag™
  Arms: relatlimab+nivolumab

SUMMARY:
This study is researching an experimental drug called fianlimab (also known as REGN3767), combined with another medication called cemiplimab (also known as REGN2810), called "study drugs". The study is focused on patients with a type of skin cancer known as melanoma. The aim of the study is to see how safe and effective the combination of fianlimab and cemiplimab is in treating melanoma, in comparison with the combination of two medications, relatlimab and nivolumab, commercialized under the brand name Opdualag™ and approved for the treatment of melanoma in adults and children.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs.
* How much study drug is in the blood at different times.
* Whether the body makes antibodies against the study drugs (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with histologically confirmed unresectable stage III and stage IV (metastatic) melanoma per American Joint Committee on Cancer (AJCC), eighth revised edition.
2. Participants must not have received prior systemic therapy for unresectable or metastatic melanoma as described in the protocol.
3. Measurable disease per RECIST version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
5. Adequate bone marrow, hepatic, and kidney function
6. Known B-Rapidly Accelerated Fibrosarcoma protein (BRAF) V600 mutation status or submitted sample for BRAF V600 mutation assessment as described in the protocol

Key Exclusion Criteria:

Medical Conditions:

1. Uveal, acral or mucosal melanoma.
2. Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents as described in the protocol.
3. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C virus (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection. Mild cancer-related immunodeficiency (such as immunodeficiency treated with gamma globulin and without chronic or recurrent infection) is allowed.

   Prior/Concomitant Therapy:
4. Prior immune checkpoint inhibitor therapy other than anti-PD1/PD-L1 as described in the protocol
5. Systemic immune suppression as described in the protocol.

   Other Comorbidities:
6. Participants with a history of myocarditis.
7. Troponin T (TnT) or troponin I (TnI) >2x institutional upper limit of normal (ULN).
8. Active or untreated brain metastases or spinal cord compression as described in the protocol.

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2033-07-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 based on blinded independent central review (BICR) | Up to 72 months

SECONDARY OUTCOMES:
Progression free survival (PFS) RECIST version 1.1 based on BICR | Up to 72 months
Death from any cause | Up to 72 months
Overall survival (OS) | Up to 72 months
Duration of Response (DOR) by BICR | Up to 72 months
DOR by investigator assessment | Up to 72 months
Disease control rate (DCR) by BICR | Up to 72 months
DCR by investigator assessment | Up to 72 months
ORR based on investigator assessment according to RECIST version 1.1 | Up to 72 months
PFS based on investigator assessment according to RECIST version 1.1 | Up to 72 months
Incidence of treatment-emergent adverse events (TEAEs) | Up to 72 months
Incidence of serious adverse events (SAEs) | Up to 72 months
Incidence of immune-mediated adverse events (imAEs) | Up to 72 months
Occurrence of interruption of study drug(s) due to AEs | Up to 72 months
Occurrence of discontinuation of study drug(s) due to AEs | Up to 72 months
TEAEs leading to death | Up to 72 months
Incidence of laboratory abnormalities | Up to 72 months
  Grade ≥3 per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) including standard hematology, chemistry, urinalysis, and other lab tests
Concentration of fianlimab in serum | Up to 72 months
Concentration of cemiplimab in serum | Up to 72 months
Incidence of anti-drug antibodies (ADAs) to fianlimab | Up to 72 months
Titer of ADAs to fianlimab | Up to 72 months
Incidence of ADAs to cemiplimab | Up to 72 months
Titer of ADAs to cemiplimab | Up to 72 months
Incidence of neutralizing antibodies (NAbs) to fianlimab | Up to 72 months
Incidence of NAbs to cemiplimab | Up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (101):
- United States (97):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Medical Foundation, Fullerton, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of California Los Angeles, Los Angeles, California
  - St. Joseph Hospital Orange, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sutter Health, Sacramento, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - St John's Cancer Institute, Santa Monica, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - The Melanoma And Skin Cancer Institute, Englewood, Colorado
  - UCHealth, Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Clermont Oncology Center, Clermont, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cancer Specialist of North Florida, Jacksonville, Florida
  - Boca Raton Clinical Research (BRCR) Global, Tamarac, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Beacon Clinic, Coeur d'Alene, Idaho
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Markey Cancer Center Clinical Research Organization, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A, Fridley, Minnesota
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - VA St. Louis Healthcare System, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Mercy South, St Louis, Missouri
  - St. Vincent Healthcare, Billings, Montana
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital Inc., Paramus, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Weisiger Cancer Institute - Charlotte, Charlotte, North Carolina
  - Duke Health System, Durham, North Carolina
  - Novant Health Zimmer Cancer Institute - Wilmington, Wilmington, North Carolina
  - Oncology Hematology Care Clinical Trials, Cincinnati, Ohio
  - Seidman Cancer Center, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Oncology Associates of Oregon PC, Eugene, Oregon
  - Kaiser Foundation Hospitals, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute (SCRI) Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Midtown Medical Center I, Austin, Texas
  - Texas Oncology - Austin Central, Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Medical City, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Center For Disease And Blood Disorder, Fort Worth, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Grapevine, Grapevine, Texas
  - Texas Oncology - Harlingen, Medical Arts Pavillion, Harlingen, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Longview, Longview, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology-Palestine Cancer Center, Palestine, Texas
  - The University of Texas Health Science Center at Tyler D/B/A UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Texas Oncology-Tyler, Northeast Texas Cancer Institute, Tyler, Texas
  - Texas Oncology - Weslaco, Knapp Medical Plaza, Weslaco, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Swedish Cancer Institute - Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute - Issaquah Campus, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Canada (4):
  - London Regional Cancer Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec (CHUQ) - Centre Hospitalier de l'Universite Laval (CHUL), Québec

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf.
URL: https://vivli.org/

REFERENCES:
- See also: Study Informational Website — https://harmonyheadtohead.com